CLINICAL TRIAL: NCT00725413
Title: A Study to Investigate the Contraceptive Efficacy and Safety of a Subdermal Etonogestrel Implant (Implanon®)
Brief Title: A Study to Investigate the Contraceptive Efficacy and Safety of a Subdermal Etonogestrel Implant (Implanon®)(P06473)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P06473; E-1729
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Healthy premenopausal women requiring a long-term method of contraception
  Interventions: Drug: etonogestrel implant (Implanon)

INTERVENTIONS:
Drug: etonogestrel implant (Implanon) — subdermal etonogestrel implant
  Other Names: Org 3236

SUMMARY:
The primary purpose of this study is to investigate the contraceptive efficacy, safety and acceptability of Organon's subdermal etonogestrel implant in healthy female volunteers in various countries in order to obtain country-specific data.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects are healthy premenopausal women requiring a long-term method of contraception, with a body mass index between 18 and 29 kg/m2, who are willing to give voluntary written informed consent. Subjects must have regular cycles with a usual length between 24 and 35 days.

Exclusion Criteria:

* Male
* Postmenopause
* Infertile
* Under 18; Over 40

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2001-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Pregnancy | Continuous, recorded at visits conducted every 3 months for the entire trial duration of 3 years.
(Serious) adverse events | Continuous, recorded at visits conducted every 3 months for the entire trial duration of 3 years.

SECONDARY OUTCOMES:
Acceptability (satisfaction questionnaire) | Every 3 months, for the entire duration of the trial